CLINICAL TRIAL: NCT01502813
Title: Citicoline, Creatine, and Omega-3 Effects in Middle Age Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Yurgelun-Todd (Other)
Responsible Party: Sponsor-Investigator, Deborah Yurgelun-Todd, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_48136
Record Dates: First submitted 2011-12-20; First posted 2012-01-02 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Benefits
Keywords: Neuropsychological testing; Dietary supplements
MeSH Terms: interventions — Cytidine Diphosphate Choline; Fatty Acids, Omega-3; Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Citicoline, Creatine, and Omega-3 Arm (Experimental): Each participant will be given a supplement log at the end of visit 1. They will be asked to complete the log during the 28 days to indicate that the daily dose of supplements were taken according to instructions. The study coordinator will check the log on the second and third visits as well as count the remaining supplement pills. If participants do not comply with the daily supplement schedule, then the PI will determine if the participant should be withdrawn from the study.
  Interventions: Drug: Citicoline, Omega-3 Fatty Acids and Creatine

INTERVENTIONS:
Drug: Citicoline, Omega-3 Fatty Acids and Creatine — Citicoline: 500 mg/day for 28 days Omega-3 Fatty Acids: 2 g/day for 28 days Creatine: 5 g/day for 28 days
  Other Names: CDP-Citicoline; Creatine monohydrate

SUMMARY:
The purpose of this study is to determine the functional effects of a citicoline, creatine, and omega-3 fatty acids combination when administered for a duration of four weeks (28 days) to non-psychiatric adult female participants.

DETAILED DESCRIPTION:
Standard clinical measures for mood and neuropsychological measures of attention, cognitive inhibition and memory will be applied before, during, and after a course of a daily supplementation of citicoline, creatine and omega-3 for 28 days to non-psychiatric adult female participants. We hypothesis that the combination of supplements will improve memory and attention in healthy adult women.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 40-60 years

Exclusion Criteria:

* Significant medical condition
* History of co-morbid psychiatric disorders
* Current Axis I or II diagnosis
* Past participation in a pharmacotherapeutic trial
* Head injury with LOC>5 minutes
* Use of psychotropic medication
* History of fish allergies
* Medical condition associated with clinically significant decreases in coagulability
* Use of anticoagulant medication

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Yurgelun-Todd, PhD, Principal Investigator — The Brain Institute, University of Utah
Locations (1):
- The Brain Institute, Salt Lake City, Utah, United States

REFERENCES:
- See also: Click here for more information about Citicoline — http://cognizin.com
- See also: Click here for more information about Omega-3 Fatty Acids — http://www.omegabrite.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Citicoline, Creatine, and Omega-3 Arm
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Forty healthy females ranging from 40 to 60 years of age (mean=48.3 ± 5.2) participated in the study.
Arm/Group | Citicoline, Creatine, and Omega-3 Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 40
Region of Enrollment [Number; unit: participants]
  United States | 40
Analyzed participants [Count of Participants; unit: Participants] | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in California Verbal Learning Test (CVLT) That Measure Attention and Memory at 14 Days
Description: List B in the California Verbal Learning Test (CVLT) score range 1-16; the score is the number of words recalled so higher scores = better performance/more words recalled.
Time Frame: Baseline and 14 days from baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Citicoline, Creatine, and Omega-3 Arm
Number analyzed (Participants) | 40
score on a scale | 10 [1 to 16]

2. Primary Outcome: Change From Baseline in WAIS-IV Block Design Subtest A That Measures Attention and Memory at 28 Days
Description: WAIS-IV Block Design Subtest A test of visuoconstructional ability is recognized as a test of visuospatial planning and function. It has been shown to be correlated with measures of general intellectual ability. The score range for this measure is 0-129. A score of 90-110 is average for a standard score. The higher the score the better the outcome.
Time Frame: Baseline and 28 days from baseline
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Citicoline, Creatine, and Omega-3 Arm
Number analyzed (Participants) | 40
Score on a scale | 98 [0 to 130]

ADVERSE EVENTS:
Time Frame: Participants were monitored for the functional effects of citicoline, creatine and omega-3 fatty acids in combination when administered for a duration of four weeks (28 days) at a daily dosage to non-psychiatric adult female subjects. The doses of 500 mg of citicoline, 5 grams of creatine, and 2 grams of omega-3 fatty acids have been selected from previous investigations and have demonstrated minimal side effects.
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Citicoline, Creatine, and Omega-3 Arm
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT01502813/Prot_SAP_000.pdf